CLINICAL TRIAL: NCT05781659
Title: The Effectiveness and Safety of Ultrasound Elastography Guided Pleural Biopsy in the Differential Diagnosis of Benign and Malignant Pleural Effusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-NHLHCRF-LX-01-0201-04
Record Dates: First submitted 2023-02-24; First posted 2023-03-23 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Pleural Effusion
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound elastography guided pleural biopsy group (Experimental)
  Interventions: Procedure: Ultrasound elastography guided pleural biopsy
- Traditional ultrasound-guided pleural biopsy group (Experimental)
  Interventions: Procedure: Traditional ultrasound guided pleural biopsy

INTERVENTIONS:
Procedure: Ultrasound elastography guided pleural biopsy — The patients will undergo ultrasound elastography (Aixplorer V, SuperSonic Imagine, FRA) guided pleural biopsy.
  Arms: Ultrasound elastography guided pleural biopsy group
Procedure: Traditional ultrasound guided pleural biopsy — The patients will undergo traditional ultrasound (Aixplorer V, SuperSonic Imagine, FRA) guided pleural biopsy.
  Arms: Traditional ultrasound-guided pleural biopsy group

SUMMARY:
The goal of this clinical trial is to evaluate the diagnostic effcacy and safety of ultrasound elastography guided pleural biopsy in the differential diagnosis of benign and malignant pleural effusion. The main question it aims to answer are: the effectiveness and safety of ultrasound elastography guided pleural biopsy in the differential diagnosis of benign and malignant pleural effusion.

Participants will undergo ultrasound elastography guided pleural biopsy or traditional ultrasound-guided pleural biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unexplained pleural effusion (patients with pleural effusion with negative aspiration)
2. Sign the informed consent form
3. The patient must have chest CT, biochemical examination of pleural fluid, cytological examination of pleural fluid and other data before operation

Exclusion Criteria:

1. The cytological examination of pleural fluid indicates "highly suspicious" patients (unless the cytological examination results of patients are inconsistent with clinical manifestations and CT examination). The pleural fluid cytology proved to be malignant. Patients with severe pleural adhesion who cannot undergo medical thoracoscopic examination will not be randomly selected, and elastic ultrasound-guided biopsy can be performed after informed consent, as a subgroup of population analysis. Those who cannot tolerate closed pleural biopsy due to severe cardiopulmonary dysfunction and poor general condition Coagulation dysfunction. Leakage. The age is less than 18 years old.
2. The pleural fluid cytology proved to be malignant.
3. Patients with severe pleural adhesion who cannot undergo medical thoracoscopic examination will not be randomly selected, and elastic ultrasound-guided biopsy can be performed after informed consent, as a subgroup of population analysis.
4. Those who cannot tolerate closed pleural biopsy due to severe cardiopulmonary dysfunction and poor general condition
5. Coagulation dysfunction.
6. transudate
7. The age is less than 18 years old.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2024-12-24 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of ultrasound elastography guided pleural biopsy versus traditional ultrasound-guided pleural biopsy for diagnosis of pleural effusion. | 7 days after the biopsy
  The diagnosis would be confirmed according to the pathological results.

SECONDARY OUTCOMES:
Incidence rate of adverse events | 7 days after the biopsy
  Symptoms and signs

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Anhui Chest Hospital, Hefei, Anhui
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Gui Zhou Provincial People's Hospital, Guiyang, Guizhou
  - the Second Xiangya Hospital of Central South University, Changsha, Hunan
  - the First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - the First Hospital of China Medical University, Shenyang, Liaoning
  - The Tenth People's Hospital of Shenyang, Shenyang, Liaoning
  - the First People's Hospital of Yunnan Provience, Kunming, Yunnan
  - the Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Deng M, Xia Y, Ye X, Ma J, Zhao S, Zhang Q, Li J, Lin J, Jing A, Li ZY, Jiang B, Wu J, Wen Q, Ma J, Tong R, Zheng Z, Xu W, Li X, Herth FJF, Hou G. Ultrasonic elastography-guided pleural biopsy versus traditional thoracic ultrasound-guided pleural biopsy for the diagnosis of pleural effusion: a multicentre, randomised trial. Eur Respir J. 2025 Dec 18;66(6):2501062. doi: 10.1183/13993003.01062-2025. Print 2025 Dec. PMID 40935584